CLINICAL TRIAL: NCT01464216
Title: MRI for Assessment of Hypoxia-Induced Prostate Cancer Aggressiveness
Acronym: FuncProst
Status: Active, not recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Therese Seierstad, Head of Research, Department of Radiology and Nuclear Medicine, Oslo University Hospital
Other Study IDs: REK-2010/1656
Record Dates: First submitted 2011-10-31; First posted 2011-11-03 (Estimated); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Prostatic Neoplasms; Genital Neoplasms, Male; Prostatic Diseases
Keywords: Functional Magnetic Resonance Imaging; Prostate cancer; FACBC PET; Hypoxia imaging
MeSH Terms: conditions — Prostatic Neoplasms; Genital Neoplasms, Male; Prostatic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, bone marrow, lymph nodes, prostate tissue, urine
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to combine and correlate data from morphological and functional MRI, molecular signatures of tumor hypoxia, the presence of micrometastases and tumor hypoxia with the goal being predicting of prostate cancer aggressiveness.

DETAILED DESCRIPTION:
A prospective study including 180 consecutive patients with PCa referred to Oslo University Hospital, Radiumhospitalet, for surgical treatment. In vivo functional MRI examination will be performed within a few days prior to robot-assisted radical prostatectomy (RALP). For a subgroup of patients FACBC PET will also be acquired prior to prostatectomy. A subgroup of intermediate and high-risk patients (D'Amico risk classification) will prior to surgery receive an intravenous infusion of the hypoxia-marker pimonidazole (Hypoxyprobe™-1)*. During surgery, bone marrow aspiration and blood collection will be performed for assessment of disseminated and circulating tumor cells. High-risk patients will undergo intraoperative lymph node dissection. Tumor tissue for molecular analyses will be sampled from prostate specimen prior to fixation. Prostate specimen and regional lymph nodes will be histopathologically examined for T- and N-classification, Gleason grade, presence of micrometastasis and areas of hypoxia. Histological and molecular findings will be correlated to MRI and PET findings and clinical data. Patients will be longitudinally followed to assess long-time clinical outcome (recurrence, metastatic disease, death).

*From 2013 oral administration is used.

ELIGIBILITY:
Inclusion Criteria:

* Patients suitable for surgery with confirmed prostate cancer, Gleason grade ≥ 3
* Patient has received no prior treatment for prostate cancer.
* Patient has adequate renal function: Estimated creatinine clearance ≥ 60 ml/minute.
* Patient must sign written informed consent according to the protocol approved by the Regional Ethics Committee.

Exclusion Criteria:

* Patient with contraindication to MR or MR contrast media according to clinical practice.
* Patients who want to withdraw for any reason during the study.
* Patients previously undergone pelvic surgery or radiation therapy

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Prostate cancer patients referred for surgical treatment.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2011-10; Primary Completion 2022-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Death | 2030

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Norway